CLINICAL TRIAL: NCT01529762
Title: A Prospective, Observational Study of Immediate Loading Cases Using Osseotite Certain Tapered Implants
Brief Title: Observational Study of Osseotite Certain Tapered Implants in Immediate Loading Cases
Acronym: Carrera
Status: Completed | Type: Observational
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Other Study IDs: 3007
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Partial Edentulism; Tooth Disease
Keywords: edentulism; dental implants; Osseotite Certain Tapered; randomized; clinical study; partial edentulism; immediate loading; crestal bone level
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Osseotite Certain Tapered: Dental implant Osseotite Certain Tapered design

SUMMARY:
Osseotite Certain Tapered implants placed in immediate prosthesis loaded cases.

DETAILED DESCRIPTION:
Osseotite Certain Tapered implants are placed and restored immediately (during the same visit)

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex and older than 18 years of age
* patients needing at least one dental implant to treat partial edentulism
* patients physically able to tolerate surgical and restorative dental procedures
* patients agreeing to all protocol visits

Exclusion Criteria:

* patients with infection or severe inflammation at the intended treatment sites
* patients smoking greater than 10 cigarettes per day
* patients with uncontrolled diabetes mellitus
* patients with uncontrolled metabolic diseases
* patients who received radiation treatment to the head in the past 12 months
* patients needing bone grafting at the intended treatment sites
* patients known to be pregnant at screening visit
* patients with para-functional habits like bruxing and clenching

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with partial edentulism needing a minimum of one dental implant restored immediately (same visit)
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2011-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
cumulative success rate | 3 years
  An implant will be considered successful if it is immobile at various study points in time

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Fuentes, DDS, Principal Investigator — Universidad San Sebastian
Locations (1):
- Universidad San Sebastian, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No